CLINICAL TRIAL: NCT02458287
Title: A 12 Week, Phase 3, Double-blind, Randomized, Placebo-controlled, Parallel Group Study To Assess The Efficacy, Safety, Tolerability And Actual Use Of Bococizumab And An Autoinjector (Pre-filled Pen) In Subjects With Primary Hyperlipidemia Or Mixed Dyslipidemia
Brief Title: Efficacy, Safety, Tolerability And Actual Use Study Of Bococizumab And An Autoinjector (Pre-Filled Pen) In Subjects With Hyperlipidemia Or Dyslipidemia
Acronym: SPIRE-AI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1481046; SPIRE-AI (Other: Alias Study Number)
Record Dates: First submitted 2015-04-02; First posted 2015-06-01 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Hyperlipidemia
Keywords: mixed dyslipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bococizumab 150mg (Experimental): Bococizumab 150mg autoinjector (pre-filled pen)
  Interventions: Biological: Bococizumab 150mg
- Bococizumab 75mg (Experimental): Bococizumab 75mg autoinjector (pre-filled pen)
  Interventions: Biological: Bococizumab 75mg
- Bococizumab 150mg placebo (Placebo Comparator): Bococizumab 150mg placebo autoinjector (pre-filled pen)
  Interventions: Biological: Bococizumab 150mg placebo
- Bococizumab 75mg placebo (Placebo Comparator): Bococizumab 75mg autoinjector (pre-filled pen)
  Interventions: Biological: Bococizumab 75mg placebo

INTERVENTIONS:
Biological: Bococizumab 150mg — Bococizumab autoinjector (pre-filled pen) combination Product. 150mg every 2 weeks for 10 weeks, subcutaneous injection.
  Arms: Bococizumab 150mg
Biological: Bococizumab 75mg — Bococizumab autoinjector (pre-filled pen) combination Product. 75mg every 2 weeks for 10 weeks, subcutaneous injection.
  Arms: Bococizumab 75mg
Biological: Bococizumab 150mg placebo — Bococizumab placebo autoinjector (pre-filled pen) combination Product. 150mg placebo every 2 weeks for 10 weeks, subcutaneous injection.
  Arms: Bococizumab 150mg placebo
Biological: Bococizumab 75mg placebo — Bococizumab placebo autoinjector (pre-filled pen) combination product. 75mg placebo every 2 weeks for 10 weeks, subcutaneous injection.
  Arms: Bococizumab 75mg placebo

SUMMARY:
This study is a multicenter, randomized study in subjects with high cholesterol receiving statins to assess the efficacy to lower LDL-C, the safety, tolerability and actual use of bococizumab and an autoinjector (pre-filled pen).

ELIGIBILITY:
Inclusion Criteria:

* Treated with a statin - Fasting LDL-C >=70mg/dL and triglycerides <=400mg/dL

Exclusion Criteria:

* Pregnant or breastfeeding females - Cardiovascular or cerebrovascular event or procedures during the past 90 days - Congestive heart failure NYHA class IV - Poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Radiant Research Incorporated, Chandler, Arizona
  - Clinical Trial Research, Lincoln, California
  - National Research Institute, Los Angeles, California
  - California Medical Research Associates Inc., Northridge, California
  - Northern California Research, Sacramento, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - ACRC - Cardiology, Atlantis, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - Clinical Research of Miami, Inc., Miami, Florida
  - Prestige Clinical Research Center, Inc., Miami, Florida
  - A & R Research Group LLC, Pembroke Pines, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research,LLC, Evanston, Illinois
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - Omega Clinical Research Center, Metairie, Louisiana
  - PharmQuest, Greensboro, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - PMG Research Of Charleston, Mt. Pleasant, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Heart Care Associates, P.C., Hopewell, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington

REFERENCES:
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481046&StudyName=A%2012%20Week%2C%20Phase%203%2C%20Double-blind%2C%20Randomized%2C%20Placebo-controlled%2C%20Parallel%20Group%20Study%20To%20Assess%20The%20Efficacy%2C%20Safety%2C%20Tolerability%20And%20Actual%20Use%20Of%20Bococizumab%20And%20An%20Autoinjector%20%28pre-filled%20Pen%29%20In%20Subjects%20With%20Primary%20Hyperlipidemia%20Or%20Mixed%20Dyslipidemia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Matched to Bococizumab 150 mg: Participants received single dose of placebo matched to bococizumab 150 milligram (mg) subcutaneous injection once in every 2 weeks over a period of 12 weeks. Participants were followed up to 18 weeks.
- Bococizumab 150 mg: Participants received single dose of bococizumab 150 mg subcutaneous injection once in every 2 weeks, over a period of 12 weeks. Participants were followed up to 18 weeks.
- Placebo Matched to Bococizumab 75 mg: Participants received single dose of placebo matched to bococizumab 75 mg subcutaneous injection once in every 2 weeks, over a period of 12 weeks. Participants were followed up to 18 weeks.
- Bococizumab 75 mg: Participants received single dose of bococizumab 75 mg subcutaneous injection once in every 2 weeks, over a period of 12 weeks. Participants were followed up to 18 weeks.
Period: Overall Study
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Started | 50 | 100 | 49 | 100
Completed | 50 | 96 | 46 | 97
Not Completed | 0 | 4 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 1
Not completed — Relocated Out of State | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg | Total
Number analyzed (Participants) | 50 | 100 | 49 | 100 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12) | 58.9 (11.5) | 61 (9.7) | 59.9 (10.1) | 60 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 42 | 29 | 48 | 137
  Male | 32 | 58 | 20 | 52 | 162

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline at Week 12 in Fasting Low Density Lipoprotein Cholesterol (LDL-C) Level for Bococizumab 150 mg Dose Group and Matched Placebo
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who were randomized. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg
Number analyzed (Participants) | 50 | 95
percent change | 6.2 (3.57) | -57.2 (2.57)
Statistical Analysis 1: Comparison: Placebo Matched to Bococizumab 150 mg vs Bococizumab 150 mg; LS-mean difference, associated 95% confidence intervals, and p-value are from MMRM model with fixed effects for treatment groups, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction as covariates; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures (MMRM); LS Mean Difference = -63.4, 95% CI 2-sided [-72.0 to -54.7], Standard Error of Mean 4.40

2. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 0 (Day 1)
Description: A successful injection based on PAT was an injection where the participant answered "yes" to all the three questions: "Were you able to inject your medicine?" "Has the blue bar moved across the window?" Was the medicine not flowing after needle withdrawn?"
Time Frame: Week 0 (Day 1)
Population: Full analysis set included all participants who were randomized. Data for this outcome measure was not planned to be analyzed for placebo arms, as pre-specified in protocol.
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 100
percentage of injections | 98

3. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 2
Description: as for outcome 2
Time Frame: Week 2
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 103
percentage of injections | 94.2

4. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 104
percentage of injections | 93.3

5. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 6
Description: as for outcome 2
Time Frame: Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 101
percentage of injections | 96

6. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 100
percentage of injections | 99

7. Primary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 150 mg Dose Group at Week 10
Description: as for outcome 2
Time Frame: Week 10
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Bococizumab 150 mg
Number analyzed (Participants) | 100
Number analyzed (injections) | 101
percentage of injections | 98.0

8. Secondary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Participant Assessment Tool (PAT) for Bococizumab 75 mg Dose Group and Combined Bococizumab 150 mg and 75 mg Dose Group at Week 0 (Day 1), 2, 4, 6, 8 and 10
Description: as for outcome 2
Time Frame: Week 0 (Day 1), 2, 4, 6, 8, 10
Population: as for outcome 2
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Groups:
- Bococizumab 150 mg + Bococizumab 75 mg: Participants received single dose of Bococizumab 150 mg SC injection in treatment arm Bococizumab 150 mg and Bococizumab 75 mg SC injection in treatment arm Bococizumab 75 mg, once every 2 weeks, over a period of 12 weeks. Participants were followed up to 18 weeks.
Arm/Group | Bococizumab 75 mg | Bococizumab 150 mg + Bococizumab 75 mg
Number analyzed (Participants) | 100 | 200
Number analyzed (injections) | 102 | 205
percentage of injections
  Week 0: number analyzed (injections) | 101 | 201
  Week 0 | 97.0 | 97.5
  Week 2 | 94.1 | 94.1
  Week 4: number analyzed (injections) | 101 | 205
  Week 4 | 99.0 | 96.1
  Week 6: number analyzed (injections) | 100 | 201
  Week 6 | 97.0 | 96.5
  Week 8: number analyzed (injections) | 100 | 200
  Week 8 | 100.0 | 99.5
  Week 10: number analyzed (injections) | 100 | 201
  Week 10 | 97.0 | 97.5

9. Secondary Outcome: Percentage of Injections That Met the Definition for Successful Assessment Using the Observer Assessment Tool (OAT) for Bococizumab 150 mg Dose, Bococizumab 75 mg Dose Group and Combined Bococizumab 150 mg and 75 mg Dose Group at Week 0 (Day 1), 4 and 8
Description: As per the OAT, a 'successful' injection was based on observer's response for the question - "Was the administration successful?''. Observer's response being 'Yes' corresponded to a successful injection.
Time Frame: Week 0 (Day 1), 4, 8
Population: Full analysis set included all participants who were randomized. Data for this outcome measure was not planned to be analyzed for placebo arms as pre-specified in protocol.
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Groups:
- Bococizumab 150 + Bococizumab 75 mg: Participants received single dose of Bococizumab 150 mg SC injection in treatment arm Bococizumab 150 mg and Bococizumab 75 mg SC injection in treatment arm Bococizumab 75 mg, once every 2 weeks, over a period of 12 weeks. Participants were followed up to 18 weeks.
Arm/Group | Bococizumab 150 mg | Bococizumab 75 mg | Bococizumab 150 + Bococizumab 75 mg
Number analyzed (Participants) | 100 | 100 | 200
Number analyzed (injections) | 105 | 103 | 206
percentage of injections
  Week 0: number analyzed (injections) | 102 | 101 | 203
  Week 0 | 99.0 | 98.0 | 98.5
  Week 4: number analyzed (injections) | 103 | 103 | 206
  Week 4 | 93.2 | 99.0 | 96.1
  Week 8: number analyzed (injections) | 105 | 100 | 205
  Week 8 | 100.0 | 100.0 | 100.0

10. Secondary Outcome: Percent Change From Baseline at Week 12 in Fasting Low Density Lipoprotein Cholesterol (LDL-C) Level for Bococizumab 75 mg Dose Group and Matched Placebo
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo Matched to Bococizumab 75 mg: Participants received single dose of placebo matched to bococizumab 75 mg subcutaneous injection once in every 2 weeks over a period of 12 weeks. Participants were followed up to 18 weeks.
Arm/Group | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 45 | 97
percent change | 6.9 (3.74) | -36.0 (2.55)
Statistical Analysis 1: Comparison: Placebo Matched to Bococizumab 75 mg vs Bococizumab 75 mg; LS-mean differences and associated 95% confidence intervals, and p-values are from an MMRM model with fixed effects for treatment groups, visit, treatment group * visit interaction, baseline value, baseline value * visit interaction as covariates; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -43.0, 95% CI 2-sided [-51.9 to -34.0], Standard Error of Mean 4.53

11. Secondary Outcome: Percent Change From Baseline in Fasting Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 50 | 97 | 45 | 97
percent change | 3.8 (2.33) | -35.9 (1.67) | 4.7 (2.45) | -22.0 (1.66)
Statistical Analysis 1: Comparison: Placebo Matched to Bococizumab 150 mg vs Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -39.7, 95% CI 2-sided [-45.4 to -34.1], Standard Error of Mean 2.86
Statistical Analysis 2: Comparison: Placebo Matched to Bococizumab 75 mg vs Bococizumab 75 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -26.7, 95% CI 2-sided [-32.5 to -20.8], Standard Error of Mean 2.96

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 50 | 96 | 45 | 97
percent change | 4.5 (3.44) | -53.4 (2.48) | 4.3 (3.62) | -31.5 (2.46)
Statistical Analysis 1: Comparison: Placebo Matched to Bococizumab 150 mg vs Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -57.9, 95% CI 2-sided [-66.2 to -49.5], Standard Error of Mean 4.25
Statistical Analysis 2: Comparison: Placebo Matched to Bococizumab 75 mg vs Bococizumab 75 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -35.8, 95% CI 2-sided [-44.4 to -27.1], Standard Error of Mean 4.38

13. Secondary Outcome: Percent Change From Baseline in Fasting Non- High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 50 | 97 | 44 | 97
percent change | 4.1 (3.12) | -52.1 (2.24) | 4.7 (3.30) | -32.5 (2.23)
Statistical Analysis 1: Comparison: Placebo Matched to Bococizumab 150 mg vs Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -56.2, 95% CI 2-sided [-63.7 to -48.6], Standard Error of Mean 3.84
Statistical Analysis 2: Comparison: Placebo Matched to Bococizumab 75 mg vs Bococizumab 75 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -37.2, 95% CI 2-sided [-45.0 to -29.3], Standard Error of Mean 3.99

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug up to the follow up visit (up to 18 weeks), that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 18 weeks
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 50 | 100 | 49 | 100
participants
  AEs | 17 | 42 | 20 | 33
  SAEs | 0 | 2 | 3 | 2

15. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb)
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported. Participants with their ADA titer levels >=6.23 were considered as ADA positive and participants with their nAb titer level >=1.58 were considered as nAb positive.
Time Frame: Baseline up to 18 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants who received at least 1 dose of bococizumab were evaluable for this outcome measure. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Bococizumab 150 mg | Bococizumab 75 mg
Number analyzed (Participants) | 97 | 99
percentage of participants
  ADA Positive | 39.2 | 22.2
  nAb Positive | 18.6 | 11.1

16. Secondary Outcome: Plasma Concentration of Bococizumab at Week 12
Time Frame: Week 12
Population: Analysis set included all participants who received at least one dose of study medication. Participants who received at least 1 dose of Bococizumab were evaluable for this outcome measure. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Bococizumab 150 mg | Bococizumab 75 mg
Number analyzed (Participants) | 92 | 90
microgram per milliliter | 6.68 (6.169) | 2.08 (1.413)

17. Secondary Outcome: Plasma Concentration of Proprotein Convertase Subtilisin Kexin Type 9 (PCSK9) at Week 12
Description: PCSK9 is an enzyme encoded by the PCSK9 gene in humans on chromosome. It is the 9th member of the proprotein convertase family of proteins that activate other proteins.
Time Frame: Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Number analyzed (Participants) | 47 | 93 | 43 | 92
nanogram per milliliter | 297.9 (102.11) | 2835.3 (901.15) | 341.8 (102.91) | 2370.9 (1016.4)

ADVERSE EVENTS:
Time Frame: Baseline up to 18 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo Matched to Bococizumab 150 mg | Bococizumab 150 mg | Placebo Matched to Bococizumab 75 mg | Bococizumab 75 mg
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/100 | 3/49 | 2/100
Other Adverse Events (participants affected / at risk) | 4/50 | 6/100 | 6/49 | 5/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matched to Bococizumab 150 mg (N=50) | Bococizumab 150 mg (N=100) | Placebo Matched to Bococizumab 75 mg (N=49) | Bococizumab 75 mg (N=100)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matched to Bococizumab 150 mg (N=50) | Bococizumab 150 mg (N=100) | Placebo Matched to Bococizumab 75 mg (N=49) | Bococizumab 75 mg (N=100)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.